CLINICAL TRIAL: NCT01565382
Title: Evaluation of Physician Training for Interpretation of Florbetapir-PET Scans: Evaluation of Inter-reader Reliability Using Images From Subjects With a Clinical Presentation of AD or MCI
Brief Title: Evaluation of Inter-reader Reliability Using Images From Subjects With Alzheimer's Disease (AD) or Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A09
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer's Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Independent, blinded reader trainees (Experimental): Seven practicing nuclear medicine physicians with no prior training in reading scans from florbetapir-PET, or other amyloid imaging agents.
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 370MBq (10mCi), single dose (intervention for Study A05 participants, source of scans for this study)
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
Re-read of brain amyloid scans acquired in previous AV-45 clinical studies by readers trained using updated reading methodology. The scans in this study came from subjects who had Alzheimer's Disease (AD) or Mild Cognitive Impairment (MCI).

ELIGIBILITY:
Participants:

* Inclusion Criteria AD:

  * Male or female >=50 years of age
  * Meet National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) criteria for probable AD with Mini-Mental State Examination (MMSE) score of 10-24
* Inclusion Criteria MCI:

  * Male or female >=50 years of age
  * Have a Clinical Dementia Rating (CDR) of 0.5
  * MMSE >24
* Exclusion Criteria:

  * Have a history or current diagnosis of other neurologic disease
  * Have had or currently have a diagnosis of other neurodegenerative disease
  * Have participated in experimental therapy targeted to amyloid plaque

Readers:

•Private nuclear medicine physicians with no prior training in reading florbetapir-PET scans

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NO SUBJECTS WERE ENROLLED IN THIS STUDY - this study re-read 40 scans obtained from 25 mild cognitive impairment (MCI) subjects and 15 Alzheimer's Disease (AD) subjects randomly selected from Study A05 (NCT00702143).
Groups:
- A05 Florbetapir-PET Scans: Subjects who received a valid florbetapir-PET scan in Study A05 (NCT00702143)
Period: Overall Study
Arm/Group | A05 Florbetapir-PET Scans
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | A05 Florbetapir-PET Scans
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Inter-reader Agreement - Median Kappa Statistic
Description: Seven readers blinded to all clinical information using the binary read methodology (amyloid positive/negative). Simple kappa statistics were calculated for each reader versus the other 6 readers. Primary outcome measure was the median kappa of each reader versus the other 6 readers.
Time Frame: 50-60 min after injection
Population: Seven private practice nuclear medicine physicians with no prior training in reading florbetapir-PET scans each rated 40 florbetapir-PET scans (7 readers x 40 scans = 280 scan reads) as either amyloid positive or negative.
Measure: Number; unit: median kappa
Units Other Than Participants: florbetapir PET scan reads
Groups:
- A05 Florbetapir-PET Scans: Subjects who received a valid florbetapir-PET scan in Study A05(NCT00702143)
Arm/Group | A05 Florbetapir-PET Scans
Number analyzed (Participants) | 40
Number analyzed (florbetapir PET scan reads) | 280
median kappa
  Reader 1 | 0.72
  Reader 2 | 0.70
  Reader 3 | 0.25
  Reader 4 | 0.75
  Reader 5 | 0.68
  Reader 6 | 0.83
  Reader 7 | 0.68

2. Secondary Outcome: Overall Inter-reader Agreement - Fleiss' Kappa
Description: Seven readers blinded to all clinical information using the binary read methodology (amyloid positive/negative). Fleiss' kappa was calculated across all inter-reader comparisons.
Time Frame: 50-60 min after injection
Population: as for outcome 1
Measure: Number; unit: Fleiss' kappa
Units Other Than Participants: florbetapir PET scans
Arm/Group | A05 Florbetapir-PET Scans
Number analyzed (Participants) | 40
Number analyzed (florbetapir PET scans) | 280
Fleiss' kappa | 0.61

ADVERSE EVENTS:
Description: Adverse Events were not collected for this study. No subjects received florbetapir in this study. This study consisted of rereads of scans previously acquired in another clinical study (A05[NCT00702143]).
Arm/Group | A05 Florbetapir-PET Scans
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days